CLINICAL TRIAL: NCT04428736
Title: ECHO: Evaluating Cascade Communication Methods
Brief Title: Evaluating Cascade Communication Methods
Acronym: ECHO
Status: Active, not recruiting | Type: Observational
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Other Study IDs: 833635
Record Dates: First submitted 2020-05-22; First posted 2020-06-11 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: BRCA1 Mutation; BRCA2 Mutation
Keywords: BRCA1; BRCA2; Cascade testing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Disclosure Toolkit — Participants will receive a "Disclosure Toolkit" consisting of a family letter, gene information chatbot, and informational website to aid in communicating their genetic test results with at-risk relatives.

SUMMARY:
Hereditary cancer programs face challenges with respect to effective communication of genetic test results within families and uptake of genetic testing by relatives. This study aims to determine if a "disclosure toolkit" provided to the index participant (carrier of cancer risk gene mutation) contributes to sharing genetic test results with relatives, if there are preferred disclosure methods, and whether toolkit use contributes towards at-risk relatives pursuing genetic testing.

DETAILED DESCRIPTION:
The identification of a single individual with a highly penetrant cancer susceptibility gene mutation can have far reaching implications for at-risk relatives in that other family members can engage in highly informative and predictive genetic testing for cancer predisposition. Family members who carry the familial cancer gene mutation are able to receive personalized cancer risk management based upon their positive test result, while those family members who test negative can generally be downgraded to follow cancer screening guidelines for the general population, barring additional familial or personal risk factors for developing cancer. Though crucial for stratifying and managing risks for relatives, familial testing, otherwise known as cascade testing, is not always successfully implemented within and across families. On a clinical basis the proband, also known as the index mutation carrier, is generally encouraged to share results with family members in order to promote their engagement in genetic counseling and testing. Despite the provision of results and a tailored letter for family members, hereditary cancer programs routinely face challenges with respect to communication of results within families and uptake of testing by relatives. Research on family communication and cascade testing substantiates this experience as previous studies have demonstrated suboptimal uptake of cascade testing in families, despite its importance for defining and managing cancer risk (Barsevicket al,2008; Daly et al, 2016). The purpose of our research study is to determine whether the provision of multiple communication tools and platforms will improve communication between probands and at-risk relatives, and if so, which communication method is the most useful to probands in communicating their results and to relatives in coming to a decision regarding genetic counseling and testing. Through the study, probands will be provided with a three-part toolkit that includes a letter, website, and a chatbot known as "GIA" (for"Genetic Information Assistant"). Though the challenges/barriers of cascade testing are well-documented, there are scant reports of follow-up with relatives. Our study allows direct contact with family members (by way of proband consent) to assess motivations and barriers to genetic testing by family members.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older
* Proband must be carrier of a high risk cancer predisposition gene
* Relative must be established relative of respective proband participant and deemed "at-risk" for familial gene mutation and eligible genetic testing candidate as per study team determination
* Participants must be able to understand and read English
* Participants must be able to provide informed verbal or written consent

Exclusion Criteria:

* <18 years of age
* Individuals who are mutation negative for high risk cancer predisposition genes
* Individuals who are carriers of a variant of uncertain significance in any gene
* Individuals who test positive for more than 1 high risk cancer predisposition gene
* Individuals who cannot speak and read English
* Individuals who do not have any at-risk relatives (eligible for familial gene mutation testing) as per study team determination
* Major psychiatric illness or cognitive impairment that in the judgement of the study investigators or study staff would preclude study participation
* Any patients who are unable to comply with the study procedures as determined by the study investigators or study staff
* No available family members for cascade opportunity (adoption, estrangement, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be ascertained through the clinical genetics programs at Penn Medicine (Mariann and Robert MacDonald Cancer Risk Evaluation Program, "CREP," the Gastrointestinal Cancer Risk Evaluation Program, "GI CREP," and Penn Telegenetics). Participants will be clinical patients identified to be a carrier of a high risk cancer predisposition gene mutation as determined by the study team. Participants will have been through a formal pre-test genetic counseling consultation and will be approached for study enrollment at time of result disclosure (either telephone or in-person) - also known as the "post-test" visit. Disclosure of genetic test results will be facilitated by a participating genetic counselor.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-02-19 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Impact of Toolkit use on sharing genetic test results with at-risk relatives | 1 year
  Determine if a "Disclosure Toolkit" contributes to participant sharing of genetic test result with at-risk relatives, and if so, which method is most useful for aiding in communication of results and decisions to undergo genetic counseling and testing.
Impact of Toolkit use on at-risk relatives pursuing genetic testing | 1 year
  Determine if a "Disclosure Toolkit" impacts the rate of genetic testing by at-risk relatives in comparison to rates of genetic testing by relatives consistently reported in the literature.

SECONDARY OUTCOMES:
Barriers to sharing genetic test results with at-risk relatives | 1 year
  Assess possible barriers and/or unforeseen challenges that inhibit optimal sharing of genetic test results with at-risk relatives.
Barriers inhibiting uptake of genetic testing by informed at-risk relatives | 1 year
  Assess possible barriers and/or unforeseen challenges that inhibit optimal uptake of genetic testing by informed at-risk relatives.

CONTACTS AND LOCATIONS:
Overall Officials: Susan M Domchek, MD, Principal Investigator — Penn Medicine
Locations (1):
- Abramson Cancer Center, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided